CLINICAL TRIAL: NCT00327236
Title: Killer T Cell Activity in the Paraneoplastic Neurologic Syndromes
Brief Title: The Study of Immune Cell (T Cell) Activity in Patients With Paraneoplastic Neurologic Syndromes
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: RDA-0148
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Paraneoplastic Syndromes
Keywords: Paraneoplastic Neurologic Syndromes
MeSH Terms: conditions — Paraneoplastic Syndromes; Paraneoplastic Syndromes, Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, cells)
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators believe that T cells, cells that are a part of the immune system, are what are causing the neurological problems while also attacking tumor cells. This protocol studies the clinical status of patients with paraneoplastic neurological disorder (PND) as well as their blood to understand the relationship between their neurological disease, their cancer, and their immune system.

DETAILED DESCRIPTION:
Patients with paraneoplastic neurological disorders (PNDs) provide a unique model for studying tumor immunity and neuronal autoimmunity. We hypothesize that T lymphocyte autoimmune dysfunction is involved in the pathogenesis of the paraneoplastic neurological syndromes, and that killer T cells are involved in the targeting and successful killing of tumor cells in these cancer patients. Furthermore, we postulate that this activity may provide a model for autoimmune brain disease. We will assess the immune responses in PND patients, correlate these with the clinical data (time course of disease, symptoms and signs, disability), and collect and archive clinical data, serum and cells from PND patients for current and future studies into the basic immune system phenomenon present in PND patients.

ELIGIBILITY:
Inclusion Criteria:

* Neurological disease which is suspected to be paraneoplastic
* No known active additional malignancy other than non-melanoma skin cancer

Exclusion Criteria:

* Known central nervous system (CNS) metastasis
* Known active additional malignancy
* No pulmonary disease which limits daily activities

if leukapheresis: must be 14 or older no known hepatitis B or C, HIV, or syphilis (by history or prior negative tests) no known IV drug users HgB > 8.5 WBC > 3,500 platelets > 100,000 INR < 2

if large blood draw (1/2 to 1 unit; children 3 ml/kg) in lieu of leukapheresis: no known IV drug users HgB > 10 WBC > 3,500 platelets > 100,000 INR < 2

if lumbar puncture: platelets > 120,000 INR < 1.2 must be 14 or older

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with paraneoplastic neurologic disease, diagnosed through the research lab of the PI, or from third party referrals in the NYC area.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 1995-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Immunologic responses to tumor antigens in vitro | throughout study
  ELISPOT

CONTACTS AND LOCATIONS:
Overall Officials: Robert Darnell, MD, PHD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States